CLINICAL TRIAL: NCT07330674
Title: A Phase 1, Single Ascending Dose and Multiple Ascending Dose Study to Assess Safety, Tolerability, and Pharmacokinetics of Orally Administered ABF- 101
Brief Title: A Phase 1 Study of ABF-101 in Single- and Multiple-Ascending Doses
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Aptabio Therapeutics, Inc. (Individual)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ABF-101-01
Record Dates: First submitted 2025-11-14; First posted 2026-01-09 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Age Related Macular Degeneration (ARMD); AMD - Age-Related Macular Degeneration
Keywords: ABF-101; AMD; NOX
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part A (ABF-101 or Placebo) (Experimental): * Part A (Phase 1a) will be a randomized, double-blind, placebo-controlled, single ascending dose (SAD) study in healthy participants.
  * Capsule, single oral dose
  Interventions: Drug: ABF-101; Drug: Placebo
- Part B (ABF-101 or Placebo) (Experimental): * Part B (Phase 1b) will be a randomized, double-blind, placebo-controlled, multiple ascending dose (MAD) study in healthy participants.
  * Capsule, once daily by mouth
  Interventions: Drug: ABF-101; Drug: Placebo
- Part C (ABF-101) (Experimental): * Part C will be an open-label study in participants with AMD
  * Capsule, once daily by mouth
  Interventions: Drug: ABF-101

INTERVENTIONS:
Drug: ABF-101 — orally, QD
Drug: Placebo — orally, QD
  Arms: Part A (ABF-101 or Placebo); Part B (ABF-101 or Placebo)

SUMMARY:
This is a Phase 1 study to evaluate the safety, tolerability, PK, and PD of ABF-101 in healthy participants and participants with age-related macular degeneration (AMD).

DETAILED DESCRIPTION:
Part A will be a randomized, double-blind, placebo-controlled, single ascending dose (SAD) study in healthy participants.

Part B will be a randomized, double-blind, placebo-controlled, multiple ascending doses (MAD) study in healthy participants.

Part C will be an open-label study in participants with AMD. For Part A and B, serial blood samples will be collected to assess the PK of ABF-101. Ocular examinations will be conducted to evaluate changes in ocular characteristics and function.

ELIGIBILITY:
Inclusion Criteria:

* Part A and B

  1. Healthy participants, aged between 18 and 50 years
  2. Provides written, signed, informed consent prior to selection
  3. BMI of ≥ 18.0 and < 32.0 kg/m2, and body weight between 50 kg and 115 kg, inclusive.
  4. Vital signs: normal pulse rate and blood pressure.
  5. Nonsmoker
  6. Must be willing to abstain from caffeine and alcohol
  7. Must be willing to avoid strenuous activity
* Part C

  1. Confirmed diagnosis of AMD
  2. Male or female ≥50 years of age
  3. Adequate visual acuity in the non-study eye

Exclusion Criteria:

* Part A and B

  1. Any history or presence of cardiovascular, pulmonary, gastrointestinal, hepatic, renal, metabolic, hematological, neurologic, psychiatric, systemic, or infectious disease
  2. Any significant abnormalities detected during ocular examination,
  3. Presence or history of drug hypersensitivity, or allergic disease diagnosed and treated by a physician
  4. Any drug intake (except paracetamol or contraceptives)
  5. History or presence alcohol abuse
  6. History or presence of drug abuse
  7. Positive HBsAg or anti-HCV antibody, or positive results for HIV
  8. Blood donation, significant blood loss, or has received a transfusion of any blood or blood products
  9. Female participants who are breastfeeding.
  10. Female participants must not be pregnant or at risk to become pregnant during the study. Male and female participants must agree to use highly effective contraception
  11. Participant who, in the judgment of the Investigator, is likely to be non-compliant or uncooperative during the study, or unable to cooperate because of a language barrier or poor mental development

Part C

1. Evidence of CNV due to any cause other than AMD
2. History of vitreoretinal surgery
3. Significant ocular diseases that may interfere with the study
4. Significantly impaired renal or hepatic function
5. Use of immunosuppressive drugs
6. Use of any investigational agent or participation in any other clinical trial of an investigational agent or investigational therapy
7. History of severe drug allergies or drug hypersensitivity syndrome
8. Undiagnosed acute illness first observed during screening or between screening and baseline, or severe concurrent medical conditions that, in the investigator's judgment, represent a safety concern.
9. Severe cardiac disease.
10. QTc ≥450 msec or participants with a history of risk factors or other clinically significant ECG abnormalities
11. Stroke or transient ischemic attack
12. Any major surgical procedure w
13. Serious active infection, other serious medical condition or any other condition that would impair the ability of the participant to administer the investigational drug or to adhere to the study protocol requirements
14. Presence of any condition which, in the judgment of the investigator, would prevent the participant from completing the study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-11 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with treatment-emergent adverse event | From enrollment up to 12 weeks
  To investigate the safety and tolerability of single ascending dose of ABF-101orally administered in healthy participants (Part A and B) and in AMD (Part C)

SECONDARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of ABF-101 | From enrollment up to 12 weeks
  Assessment of the maximum observed plasma concentration
Time to maximal concentration (Tmax) of ABF-101 | From enrollment up to 12 weeks
  Assessment of time to maximal concentration
The plasma area under the curve (AUC) of ABF-101 | From enrollment up to 12 weeks
  Assessment of the plasma area under the curve
Terminal elimination half-life of ABF-101 | From enrollment up to 12 weeks
  Assessment of terminal elimination half-life

CONTACTS AND LOCATIONS:
Locations (1):
- Dallas Clinical Research Unit, Dallas, Texas, United States